CLINICAL TRIAL: NCT01778374
Title: Mater _Bronx Rapid HIV Testing Project. Prospective Randomised Trial of Recruitment Methods in Implementation of a HIV Screening Programme in the Emergency Department.
Brief Title: Mater-Bronx Rapid HIV Testing Project.
Acronym: M-BRiHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Patrick Mallon, Associate Dean for Research and Innovation UCD School of Medicine and Medical Sciences, Consultant Infectious Diseases Physician, Head of HIV Molecular Research Group (HMRG)., University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: M-BRiHT
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: Emergency Medicine; Screening; Point of care testing; Video assisted counseling
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No participant choice of counselor (Experimental): Participants in this arm of the study are randomized to an interactive video counselor with no choice of counselor. This is delivered via a touchscreen tablet device.
  Interventions: Other: No participant choice of counselor
- Participant choice of counselor (Experimental): Participants in this arm of the study are randomized to an interactive video counselor with a choice of four different counselors. These gender and ethnically diverse counselors are delivered via a touchscreen tablet device.
  Interventions: Other: Participant choice of counselor

INTERVENTIONS:
Other: No participant choice of counselor — Participants in this arm of the study are randomized to an interactive video counselor with no choice of counselor. This is delivered via a touchscreen tablet device.
  Arms: No participant choice of counselor
Other: Participant choice of counselor — Participants in this arm of the study are randomized to an interactive video counselor with a choice of four different counselors. These gender and ethnically diverse counselors are delivered via a touchscreen tablet device.
  Arms: Participant choice of counselor

SUMMARY:
In the M-BRiHT study we aim to implement a programme of opportunistic HIV screening in the Emergency Department, Mater Misericordiae University Hospital. We hypothesize that such a programme will be acceptable in an Irish setting. We also wish to study the factors that influence test completion or acceptance. We will utilise informative interactive video media via a touch-screen tablet device to provide pre-test counselling and then offer rapid minimally invasive testing with a cotton-bud type swab of the buccal mucosa. In doing so we will to determine absolute numbers of those attending the ED who consent to watching the interactive information video about rapid HIV test screening. We will describe the absolute number and proportion of those who watch the interactive video who subsequently proceed to have the rapid HIV test. The primary aim is to determine the cultural, gender and ethnic factors which influence the completion of such rapid HIV testing with the future objective of maximising test completion in this crucial public health area.

ELIGIBILITY:
Inclusion Criteria:

* All adults greater than 18 years of age who present to the Emergency Department, Mater Misericordiae University Hospital
* Must have capacity to consent to watch an interactive video tablet device about HIV and HIV screening test.

Exclusion Criteria:

* HIV positive patients (known previous HIV positive patients).
* Acute intoxication in which capacity is impaired
* Critically unwell patients who require active or intensive resuscitation.
* Acute psychiatric disturbance in which capacity is impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17000 (Estimated)
Dates: Start 2012-09; Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients agreeing to undergo a HIV screening test in the Emergency Department | 24 months
  Establish a programme of HIV screening in the Emergency Department, Mater Misericordiae University Hospital. Acceptability of the programme will be judged in terms of absolute numbers of patients consenting to the test.

SECONDARY OUTCOMES:
To determine the proportions of those who test negative who may fall in to the three month seroconversion window and to determine the proportion of those who return for repeat/multiple HIV tests at three months or other time in the future. | 24 months
Absolute numbers of those attending the ED who consent to watching the interactive information video about rapid HIV test screening. | 24 months
Absolute number and proportion of HIV positive test results | 24 months
CD4 count and viral load of newly diagnosed HIV positive patients | 24 months
Number of those testing positive who have acute seroconversion illness | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick WG Mallon, MB, BCh, BAO, FRACP, FRCPI,PhD, Principal Investigator — Group Leader, HIV Molecular Research Group, University College Dublin; Gerard S O'Connor, MB, BCh, BAO, MCEM, MMed, Study Director — Project Lead M-BRiHT, HIV Molecular Research Group, University College Dublin.; Yvette Calderon, MD, Study Director — Jacobi Medical Centre, New York
Locations (1):
- Emergency Department, Mater Misericordiae University Hospital., Dublin, Ireland

REFERENCES:
- [Background] Centers for Disease Control (CDC). Pneumocystis pneumonia--Los Angeles. MMWR Morb Mortal Wkly Rep. 1981 Jun 5;30(21):250-2. No abstract available. PMID 6265753
- [Background] Wilson JM, Jungner YG. [Principles and practice of mass screening for disease]. Bol Oficina Sanit Panam. 1968 Oct;65(4):281-393. No abstract available. Spanish. PMID 4234760
- [Background] Jacquez JA, Koopman JS, Simon CP, Longini IM Jr. Role of the primary infection in epidemics of HIV infection in gay cohorts. J Acquir Immune Defic Syndr (1988). 1994 Nov;7(11):1169-84. PMID 7932084
- [Background] Pilcher CD, Tien HC, Eron JJ Jr, Vernazza PL, Leu SY, Stewart PW, Goh LE, Cohen MS; Quest Study; Duke-UNC-Emory Acute HIV Consortium. Brief but efficient: acute HIV infection and the sexual transmission of HIV. J Infect Dis. 2004 May 15;189(10):1785-92. doi: 10.1086/386333. Epub 2004 Apr 28. PMID 15122514
- [Background] Wawer MJ, Gray RH, Sewankambo NK, Serwadda D, Li X, Laeyendecker O, Kiwanuka N, Kigozi G, Kiddugavu M, Lutalo T, Nalugoda F, Wabwire-Mangen F, Meehan MP, Quinn TC. Rates of HIV-1 transmission per coital act, by stage of HIV-1 infection, in Rakai, Uganda. J Infect Dis. 2005 May 1;191(9):1403-9. doi: 10.1086/429411. Epub 2005 Mar 30. PMID 15809897
- [Background] Chakraborty H, Sen PK, Helms RW, Vernazza PL, Fiscus SA, Eron JJ, Patterson BK, Coombs RW, Krieger JN, Cohen MS. Viral burden in genital secretions determines male-to-female sexual transmission of HIV-1: a probabilistic empiric model. AIDS. 2001 Mar 30;15(5):621-7. doi: 10.1097/00002030-200103300-00012. PMID 11317000
- [Background] Gray RH, Wawer MJ, Brookmeyer R, Sewankambo NK, Serwadda D, Wabwire-Mangen F, Lutalo T, Li X, vanCott T, Quinn TC; Rakai Project Team. Probability of HIV-1 transmission per coital act in monogamous, heterosexual, HIV-1-discordant couples in Rakai, Uganda. Lancet. 2001 Apr 14;357(9263):1149-53. doi: 10.1016/S0140-6736(00)04331-2. PMID 11323041
- [Background] Attia S, Egger M, Muller M, Zwahlen M, Low N. Sexual transmission of HIV according to viral load and antiretroviral therapy: systematic review and meta-analysis. AIDS. 2009 Jul 17;23(11):1397-404. doi: 10.1097/QAD.0b013e32832b7dca. PMID 19381076
- [Background] Daar ES, Pilcher CD, Hecht FM. Clinical presentation and diagnosis of primary HIV-1 infection. Curr Opin HIV AIDS. 2008 Jan;3(1):10-5. doi: 10.1097/COH.0b013e3282f2e295. PMID 19372938
- [Background] Schacker T, Collier AC, Hughes J, Shea T, Corey L. Clinical and epidemiologic features of primary HIV infection. Ann Intern Med. 1996 Aug 15;125(4):257-64. doi: 10.7326/0003-4819-125-4-199608150-00001. PMID 8678387
- [Background] Greenwald JL, Burstein GR, Pincus J, Branson B. A rapid review of rapid HIV antibody tests. Curr Infect Dis Rep. 2006 Mar;8(2):125-31. doi: 10.1007/s11908-006-0008-6. PMID 16524549
- [Background] Branson BM, Handsfield HH, Lampe MA, Janssen RS, Taylor AW, Lyss SB, Clark JE; Centers for Disease Control and Prevention (CDC). Revised recommendations for HIV testing of adults, adolescents, and pregnant women in health-care settings. MMWR Recomm Rep. 2006 Sep 22;55(RR-14):1-17; quiz CE1-4. PMID 16988643
- [Background] Centers for Disease Control and Prevention (CDC). Expanded HIV testing and trends in diagnoses of HIV infection - District of Columbia, 2004-2008. MMWR Morb Mortal Wkly Rep. 2010 Jun 25;59(24):737-41. PMID 20577154
- [Background] Donnell D, Baeten JM, Kiarie J, Thomas KK, Stevens W, Cohen CR, McIntyre J, Lingappa JR, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Heterosexual HIV-1 transmission after initiation of antiretroviral therapy: a prospective cohort analysis. Lancet. 2010 Jun 12;375(9731):2092-8. doi: 10.1016/S0140-6736(10)60705-2. Epub 2010 May 26. PMID 20537376
- [Background] Calderon Y, Haughey M, Leider J, Bijur PE, Gennis P, Bauman LJ. Increasing willingness to be tested for human immunodeficiency virus in the emergency department during off-hour tours: a randomized trial. Sex Transm Dis. 2007 Dec;34(12):1025-9. doi: 10.1097/OLQ.0b013e31814b96bb. PMID 18032992
- [Background] Haukoos JS, Hopkins E, Byyny RL; Denver Emergency Department HIV Testing Study Group. Patient acceptance of rapid HIV testing practices in an urban emergency department: assessment of the 2006 CDC recommendations for HIV screening in health care settings. Ann Emerg Med. 2008 Mar;51(3):303-9, 309.e1. doi: 10.1016/j.annemergmed.2007.10.028. Epub 2008 Jan 11. PMID 18191295
- [Background] Freeman AE, Sattin RW, Miller KM, Dias JK, Wilde JA. Acceptance of rapid HIV screening in a southeastern emergency department. Acad Emerg Med. 2009 Nov;16(11):1156-64. doi: 10.1111/j.1553-2712.2009.00508.x. PMID 20053236
- [Background] White DA, Scribner AN, Schulden JD, Branson BM, Heffelfinger JD. Results of a rapid HIV screening and diagnostic testing program in an urban emergency department. Ann Emerg Med. 2009 Jul;54(1):56-64. doi: 10.1016/j.annemergmed.2008.09.027. Epub 2008 Nov 5. PMID 18990468
- [Background] Torres M. Rapid HIV screening in the emergency department. Emerg Med Clin North Am. 2010 May;28(2):369-80, Table of Contents. doi: 10.1016/j.emc.2010.01.008. PMID 20413019
- [Background] Haukoos JS, Hopkins E, Conroy AA, Silverman M, Byyny RL, Eisert S, Thrun MW, Wilson ML, Hutchinson AB, Forsyth J, Johnson SC, Heffelfinger JD; Denver Emergency Department HIV Opt-Out Study Group. Routine opt-out rapid HIV screening and detection of HIV infection in emergency department patients. JAMA. 2010 Jul 21;304(3):284-92. doi: 10.1001/jama.2010.953. PMID 20639562
- [Background] Merchant RC, Clark MA, Mayer KH, Seage Iii GR, DeGruttola VG, Becker BM. Video as an effective method to deliver pretest information for rapid human immunodeficiency testing. Acad Emerg Med. 2009 Feb;16(2):124-35. doi: 10.1111/j.1553-2712.2008.00326.x. Epub 2008 Dec 18. PMID 19120050
- [Background] Evans AE, Edmundson-Drane EW, Harris KK. Computer-assisted instruction: an effective instructional method for HIV prevention education? J Adolesc Health. 2000 Apr;26(4):244-51. doi: 10.1016/s1054-139x(99)00093-2. PMID 10734271
- [Background] Fureman I, Meyers K, McLellan AT, Metzger D, Woody G. Evaluation of a video-supplement to informed consent: injection drug users and preventive HIV vaccine efficacy trials. AIDS Educ Prev. 1997 Aug;9(4):330-41. PMID 9376207
- [Background] Reznik M, Sharif I, Ozuah PO. Use of interactive videoconferencing to deliver asthma education to inner-city immigrants. J Telemed Telecare. 2004;10(2):118-20. doi: 10.1258/135763304773391585. PMID 15068650
- [Background] Calderon Y, Haughey M, Bijur PE, Leider J, Moreno-Walton L, Torres S, Gennis P, Bauman LJ. An educational HIV pretest counseling video program for off-hours testing in the emergency department. Ann Emerg Med. 2006 Jul;48(1):21-7. doi: 10.1016/j.annemergmed.2006.01.003. Epub 2006 Mar 13. PMID 16781919
- [Background] Calderon Y, Leider J, Hailpern S, Haughey M, Ghosh R, Lombardi P, Bijur P, Bauman L. A randomized control trial evaluating the educational effectiveness of a rapid HIV posttest counseling video. Sex Transm Dis. 2009 Apr;36(4):207-10. doi: 10.1097/OLQ.0b013e318191ba3f. PMID 19265735
- [Background] Calderon Y, Leider J, Hailpern S, Chin R, Ghosh R, Fettig J, Gennis P, Bijur P, Bauman L. High-volume rapid HIV testing in an urban emergency department. AIDS Patient Care STDS. 2009 Sep;23(9):749-55. doi: 10.1089/apc.2008.0270. PMID 19698029